CLINICAL TRIAL: NCT06697925
Title: Prospective Multicenter Observational Study Evaluating the Durability of Closure for Venous Leg Ulcers Following a Randomized, Controlled, Clinical Trial
Brief Title: Evaluating the Durability of Closure for Venous Leg Ulcers
Acronym: THORSDOTTIR
Status: Recruiting | Type: Observational
Sponsor: Kerecis Ltd. (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Other Study IDs: KS-1020
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Venous Leg; Venous Leg Ulcer (VLU); Venous Leg Ulcer; Venous Ulcer; VLU
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thor closure patients: Patients who achieved closure in during the THOR clinical trial

SUMMARY:
The goal of this observational study is to determine the durability of closure for venous leg ulcer subjects that achieved closure in the THOR trial.

DETAILED DESCRIPTION:
To determine durability of closure (rate of target wound recurrence) of subjects with a closed venous leg ulcer during the THOR clinical trial comparing subjects treated with Intact Fish Skin Graft (IFSG) plus standard of care (SOC) to subjects treated with SOC alone.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must have participated in the THOR trial and achieved complete closure by the 12-week endpoint.

Exclusion Criteria:

* 1. Subjects who did not participate in the THOR trial. 2. Subjects who participated in the THOR trial and did not achieve complete closure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who achieved closure in during the THOR clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Durability of closure | 12-month follow-up
  To demonstrate durability of closure (rate of target wound recurrence) of subjects with a closed venous leg ulcer during the THOR clinical trial comparing subjects treated with Intact Fish Skin Graft (IFSG) plus standard of care (SOC) to subjects treated with SOC alone.

CONTACTS AND LOCATIONS:
Locations (1):
- Serena Group, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No